CLINICAL TRIAL: NCT06687954
Title: Activation of the Ankle Musculature During the Sporting Gesture in Basketball Players With Chronic Ankle Instability A Case Control Study
Brief Title: Activation of the Ankle Musculature in Basketball Players With Chronic Ankle Instability
Status: Completed | Type: Observational
Sponsor: Camilo Jose Cela University (Other)
Responsible Party: Sponsor
Other Study IDs: 15_24_CQSI
Record Dates: First submitted 2024-11-03; First posted 2024-11-14 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Chronic Ankle Instability, CAI

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 58 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Players of basketball team without CAI: this players have no history of ankle sprain
- Case: Players of basketball team with CAI: scored ≥ 11 on the functional ankle instability identification questionnaire.

SUMMARY:
Background: Lateral ankle sprain (LAS) is a very common injury in the general population and in the world of basketball in particular, initially Its recurrence rate is very high, generating chronic ankle instability (CAI), accompanied by decreased muscle activation in the ankle musculature and lack of motor control. The aim of this study is to evaluate the activation of the peroneal musculature during the sports gestures of layup and free throw, and the motor control of both in healthy patients and in patients with CAI.

Method: Using a surface electromyography study (sEMG) of 58 basketball players of amateur teams, 36 women and 22 men, with and without CAI, in the peroneus lateralis longus (PLL) and peroneus lateralis brevis musculature (PLB).

DETAILED DESCRIPTION:
Design A case-control study was conducted. The entire procedure was carried out for human experimentation. The case control study followed the CONSORT guidelines.

Meassurement Muscle activity was recorded using an mDurance R surface EMG system (mDurance Solutions SL, Granada, Spain), a portable sEMG system that consists of three parts(i) A Shimmer3 EMG unit (Realtime Technologies Ltd., Dublin, Ireland), which is a bipolar sEMG sensor for muscle activity acquisition. Each Shimmer sensor is composed of two sEMG channels, with a sampling rate of 104 Hz. (ii) The mDurance mobile application (Android), which receives data from the Shimmer unit and sends it to a cloud service(iii) The mDurance cloud service, where the sEMG signals were stored, filtered and analysed, and reports were generated.

Surface electrode placement was performed following the recommendations of Surface EMG for Non-Invasive Muscle Assessment (SENIAM),bilaterally and parallel to the direction of the muscle fibres.

Protocol Firstly, anthropometric variables and personal information, training hours of the participants as well as ankle and lower limb injuries were collected through a Microsoft Forms.

In this study, changes in the sEMG signal of PLL and PLB in patients with and without CAI were investigated in the performance of various basketball-specific sport gestures . These changes in signal amplitude (root mean square) reflect the level of activation during the sporting gesture in the PLL and PLB muscles.

Maximal voluntary contraction (MVC) measurement First, participants were asked to perform a MVC, both PLL and PLB towards eversion and in the supine position, from the inversion position. Three maximal attempts of 5 seconds each, separated by 1 minute of rest, were performed. The best performance was chosen for statistical analysis.

Participants were verbally encouraged as the investigators conducted the assessment. The purpose of this test was to compare maximal amplitudes with submaximal amplitudes.

EMG recording in sport gesture The participants first warmed up for 10 minutes on the court, after which they were ready to shoot 3 series of 18 free throws each, with a rest of 35 seconds between each of them. The first sport gesture measured was the free throw, that is a sporting gesture that is always performed from a distance of 4.57 metres from the basket, which is 305 cm high. They were always performed with the same ball, with a perimeter size of 74.93 - 78 cm in the case of the male category and 72.4 - 73.7 cm in the case of the female category, as per National Basketball Association standards. To avoid fatigue, each shot was separated by a 10-15 second break and each series by 35 seconds. All participants in the study performed the throws without instructions or instructions on how to execute each personal routine.

This was followed by 1 series of 10 right-handed basket layups(first step starting with the right leg and second starting with the left leg) and another series of 10 left-handed basket layups (first step starting with the left leg and second starting with the right leg). In between, the players were asked to rest for 5 minutes.

The drive to the basket is a sporting gesture that consists of taking 3 steps towards the basket, (i) a short step towards the basket, (ii) a long step towards the basket, and (iii) a final jump.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers aged 18-45 years
* Physical activity level of at least 3 hours per week
* First sprain more than one year ago
* No sprain in the 6 weeks prior to the test
* Scored ≥ 11 on the functional ankle instability identification questionnaire.

Exclusion Criteria:

* Having undergone lower limb surgery and/or diseases that may influence neuromuscular control
* Suffering from any type of incapacity to complete the proposed sporting gesture
* Patients without CAI should not have a history of ankle sprains.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants were selected through non-probabilistic sampling in several amateur basketball teams in the Autonomous Community of Madrid.
  Both male and female basketball players with and without CAI were recruited A total of 58 subjects participated in the study with a mean age of 29.19±6.98 years a weight of 66,46±7,23 Kilograms and a height of 1,74±0,07 meters, with a body mass index (BMI), obtained by dividing weight by height squared (kg/m^2), average of 21.87±1.64, with no differences between the two groups.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2023-12-27 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2024-07-22 (Actual)

PRIMARY OUTCOMES:
Measurement of the different activation patron of the peroneal muscles (electromyograpic analysis), in the different phases of the layup gesture , in patients with CAI and without CAI. | Up to 28 weeks
  As a primary outcome measure, the investigators evaluated the difference in the activation of the PLL and PLB muscles both in patients suffering from CAI and in those who do not suffer from it, during the development of the layup.

SECONDARY OUTCOMES:
Evaluation of moment of greatest activation (electromyographic evaluation) of the peroneal muscles, and motor control in layup gesture, in patients with CAI and without CAI. | Up to 28 weeks
  As secondary outcome measure:
  1. To evaluate the moment of greatest solicitation of these muscles during both layup gesture in healthy patients and to assess the response of the peroneal muscles at the same moment in patients with CAI.
  2. To assess the motor control in CAI patients at the moment of greatest solicitation of the ankle and their possible response to a possible injury gesture.

CONTACTS AND LOCATIONS:
Overall Officials: María Benito, Principal Investigator — Associate Professor
Locations (1):
- Universidad Camilo Jose Cela, Villanueva de la Cañada, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
Other researchers participated by collecting data from the sample, but at no time did they have access to the personal data of said sample, only to the code that represented each of them (always coded information)